CLINICAL TRIAL: NCT06220877
Title: Efficacy of Buccal Pad of Fat, Advanced Platelet Rich Fibrin, Fibrin Glue and Oxidized Cellulose Plug in Management of Oro-Antral Communication, Comparative Clinical Study
Acronym: OAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Nermine Ramadan Mahmoud, associate professor oral and maxillofacial surgery, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECO6U/19-2020
Record Dates: First submitted 2024-01-13; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteers Only
Keywords: Benacel;; bone regeneration;; platelet rich growth factor;; Oro-Antral Communication; buccal pad of fat; fibrin glue
MeSH Terms: conditions — Oroantral Fistula | interventions — Fibrin Tissue Adhesive; Cellulose, Oxidized

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (Active Comparator): patients were treated using Buccal Pad of Fat for management of OAC.
  Interventions: Procedure: Buccal Pad of Fat
- Group II (Active Comparator): patients were treated using A-PRF technique for management of OAC.
  Interventions: Procedure: A-PRF
- Group III (Active Comparator): patients were treated with Fibrin Glue for management of OAC.
  Interventions: Procedure: fibrin glue
- Group IV (Active Comparator): oxidized regenerated cellulose plug have been used for management of OAC.
  Interventions: Procedure: oxidized cellulose

INTERVENTIONS:
Procedure: Buccal Pad of Fat — surgical procedure
  Arms: Group I
Procedure: A-PRF — blood sample
  Arms: Group II
Procedure: fibrin glue — procedure
  Arms: Group III
Procedure: oxidized cellulose — procedure
  Arms: Group IV

SUMMARY:
Evaluation of the efficacy of different treatment protocols in the management of Oro-Antral Communications.

DETAILED DESCRIPTION:
the current study was carried on 24 patients suffering from Oro-Antral Communications. All patients were divided into 4 equal groups.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from oroantral communications
* patients suffering from oroantral fistula.
* The Diameter of the opening ranged from 4-9 mm,
* communication resulted from recent extraction,
* foreign body; or
* cyst enucleation

Exclusion Criteria:

Patients suffering from any systemic diseases were excluded from the study.

* diabetes,
* autoimmune diseases,
* cancers,
* nephropathy,
* coagulation disorders

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
o Recurrence | 6 months
  presence or absence

SECONDARY OUTCOMES:
pain, visual analog scale | 4 weeks
  0 no pain, 10 severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- October 6U, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mahmoud NR. Buccal pad of fat, advanced platelet-rich fibrin, fibrin glue, and oxidized cellulose plug in the management of oroantral communication: A comparative clinical study. J Stomatol Oral Maxillofac Surg. 2025 Oct;126(5S):102376. doi: 10.1016/j.jormas.2025.102376. Epub 2025 Apr 15. PMID 40246197